CLINICAL TRIAL: NCT06847672
Title: Comparison of the Time to Reach End-Tidal Oxygen Value of 90 and Oxygen Reserve Index Decline Times During Preoxygenation in Sarcopenic and Non-Sarcopenic Patients Using the 6-Minute Walk Test
Brief Title: Comparison of the Time to Reach End-Tidal Oxygen Value of 90 and Oxygen Reserve Index Decline Times During Preoxygenation in Sarcopenic and Non-Sarcopenic Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Betül Güven, Ankara Bilkent City Hospital, Ankara City Hospital Bilkent
Other Study IDs: TABED1-25-884
Record Dates: First submitted 2025-02-18; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Sarcopenia; Preoxygenation; Oxygen Reserve Index
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- sarcopenic: sarcopenia based on the 6-minute walk test results.
  Interventions: Diagnostic Test: preoxygenation
- non-sarcopenic: non-sarcopenia based on the 6-minute walk test results.
  Interventions: Diagnostic Test: preoxygenation

INTERVENTIONS:
Diagnostic Test: preoxygenation — The time required to reach EtO2 90% and the time until ORI drops below 0.55

SUMMARY:
The purpose of this study is to compare the time required to reach an end-tidal oxygen (EtO2) value of 90% and the time until the Oxygen Reserve Index (ORI) drops below 0.55 during preoxygenation in sarcopenic and non-sarcopenic patients. The study aims to investigate the impact of sarcopenia on the oxygenation process.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree to participate in the study.
* Patients scheduled for major abdominal oncologic surgery.

Exclusion Criteria:

* Patients with severe cardiopulmonary disease.
* Patients with walking disabilities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 patients who agreed to participate in the study and are scheduled for major abdominal oncological surgery will be included in the study.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Time required to reach EtO2 90% | preoperatively
Time until ORI drops below 0.55 | preoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital Bilkent, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided